CLINICAL TRIAL: NCT04845230
Title: Fresh RX: Nourishing Healthy Starts Clinical Study
Brief Title: Fresh RX: NHS 2020
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Operation Food Search Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 202011018
Record Dates: First submitted 2021-03-29; First posted 2021-04-14 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Premature Birth; Birth Weight; Post Partum Depression; Health Care Utilization; Nutrition Deficiency Due to Insufficient Food; Housing Problems; Fetal Complications; Food Deprivation
Keywords: food insecurity; pregnancy; maternal health; neonatal health; birth outcomes; poverty; health care utilization; field experiment; integrative care
MeSH Terms: conditions — Premature Birth; Birth Weight; Depression, Postpartum; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: This is a three-arm experiment where each arm iteratively adds additional program components (see study description for more detail).
Who Masked: Outcomes Assessor
Masking Description: Blinding of participants or Operation Food Search staff is infeasible in this study. Operation Food Search will need to know participants' treatment assignment in order to provide the appropriate services, and the participants will also be aware of the services they receive from Operation Food Search. However, the administrative health care claims data used to assess outcomes in this study will not be subject to any bias, as the entities responsible for entering those claims will be blind to the treatment assignment of participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced Usual Care (Active Comparator): The control group in this study will still receive some services above and beyond the usual standard of care offered to pregnant women on Medicaid. In addition to the case management services offered through their managed care provider, Operation Food Search will offer this group access to the "hunger hotline," a service provided by Operation Food Search to help them find food assistance around St. Louis; assistance in enrolling in public nutrition assistance programs like SNAP and WIC; and guidance on food pantry access in St. Louis.
  Interventions: Behavioral: FreshRx Nourishing Healthy Starts
- Treatment 1: Nutrition Services (Experimental): This treatment group will receive all the services offered to the control group, as well as the following services:
  Weekly food deliveries of fresh food meal kits with step-by-step recipes from the time of program enrollment through 60 days post-partum. Access to necessary cooking tools for their kitchen (e.g., spatulas, cutting boards , etc.), should they need them. Access to online cooking resources to help guide them on culinary skills and recipe preparation. Nutrition education and counseling provided by a registered dietitian.
  Interventions: Behavioral: FreshRx Nourishing Healthy Starts
- Treatment 2: Integrated Care Services (Experimental): This treatment group will receive all the services offered to Treatment Group 1, as well as the services of a Licensed Masters Social Worker who will provide trauma-informed integrative care services to participants. These services will focus on an array of potential needs that may emerge in participants' lives, such as assistance in finding stable housing, assistance navigating social services, connections with other community organizations, and other needs.
  Interventions: Behavioral: FreshRx Nourishing Healthy Starts

INTERVENTIONS:
Behavioral: FreshRx Nourishing Healthy Starts — This is a field experiment study that incorporates referrals to public programs, food supplementation and nutrition education, or integrative care services provided by a Licensed Masters Social Worker.

SUMMARY:
This study is an evaluation of the Fresh Rx: Nourishing Healthy Starts program administered by Operation Food Search, a St. Louis-based nonprofit organization. The program provides food and nutrition supports to food insecure pregnant women in conjunction with integrative care services in order to improve health and birth outcomes for both the mother and the child. The purpose of this study is to test the efficacy of this approach through a field experiment, and to assess the extent to which these services can provide cost savings to the healthcare system.

DETAILED DESCRIPTION:
This study is an evaluation of the Fresh Rx: Nourishing Healthy Starts program administered by Operation Food Search, a St. Louis-based nonprofit organization. The goal of the program is to provide food and nutrition supports to food insecure pregnant women in order to improve health and birth outcomes for both the mother and the child. Specifically, this program provides:

* Facilitated access to food support programs like the Supplemental Nutrition Assistance Program (SNAP); Women, Infants, and Children (WIC); and food pantries
* Direct food delivery to pregnant women, nutrition education, and access to a registered dietitian
* Access to a social worker who will provide integrative care services

Participants in this program will be recruited through a Medicaid Managed Care Organization (MCO). During their initial intake meeting with an MCO case manager, potential participants will be screened for food insecurity through the use of a two-item food insecurity screener. If a potential participant screens positive for food insecurity, she will be referred to Operation Food Search to begin the Nourishing Healthy Starts recruitment process. Consenting participants will be randomly assigned to one of three conditions (described in detail below), each of which provides the standard of care women would receive in the absence of the program plus additional program features.

Control Group. The control group in this study will still receive some services above and beyond the usual standard of care offered to pregnant women on Medicaid. In addition to the case management services offered through their managed care provider, Operation Food Search will offer this group access to the "hunger hotline," a service provided by Operation Food Search to help them find food assistance around St. Louis; assistance in enrolling in public nutrition assistance programs like SNAP and WIC; and guidance on food pantry access in St. Louis.

Treatment 1: Food Supplementation and Education Group. This treatment group will receive all the services offered to the control group, as well as the following services:

1. Weekly food deliveries of fresh food meal kits with step-by-step recipes from the time of program enrollment through 60 days post-partum;
2. Access to necessary cooking tools for their kitchen (e.g., spatulas, cutting boards , etc.), should they need them.
3. Access to online cooking resources to help guide them on culinary skills and recipe preparation.
4. Nutrition education and counseling provided by a registered dietitian.

Treatment 2: Food Supplementation, Education, and Integrative Case Management. This treatment group will receive all the services offered to Treatment Group 1, as well as the services of a licensed social worker who will provide trauma-informed integrative care services to participants. These services will focus on an array of potential needs that may emerge in participants' lives, such as assistance in finding stable housing, assistance navigating social services, connections with other community organizations, and other needs.

This evaluation will combine longitudinal survey data from participants with health claims data provided by the MCOs. Study participants will consent to have their data collected and linked for research purposes. The research team will not have access to any personally identifiable information on program participants, and the team will analyze a deidentified dataset.

Each intervention approach will examine a different method of providing women with access to affordable, nutritious food throughout their pregnancy and through the early post-partum period. After it is determined how best to support food insecure women and their families, the evidence from this study may be used to make a case for treating healthy food supports as part of a new standard of care for food insecure pregnant women. The results will provide information to public health agencies, public insurance systems, Medicaid MCOs, and other insurance companies in order to help them understand the potential benefits of these food supports.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Pregnant
* Less than 24 weeks gestation
* Screening positive to a USDA two-item food insecurity screener (described below)
* Receiving care through a Missouri Medicaid managed care organization
* English speaking
* Age 14-55
* Missouri resident residing in the following zip codes: 63031, 63033, 63042, 63074, 63114, 63121, 63130, 63132, 63133, 63135, 63136, 63137, 63138, 63140

Exclusion Criteria:

* Male
* Non-pregnant
* Pregnant, but more than 24 weeks gestation
* Does not screen positive to a USDA two-item food insecurity screener (described below)
* Does not receive care through the Home State Health managed care organization
* Non-English speaking
* Aged less than 14 or more than 55
* Does not reside in the following zip codes: 63031, 63033, 63042, 63074, 63114, 63121, 63130, 63132, 63133, 63135, 63136, 63137, 63138, 63140

Ages: 14 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — This study is an evaluation of a program that provides food and nutrition supports to food insecure pregnant women.
Enrollment: 750 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in food insecurity | Baseline, around 3 months post-baseline, 60 days post-partum, one year post-partum
  Repeated measures of food insecurity using United States Department of Agriculture (USDA) food insecurity screener
Gestational Age at Birth | Collected at time of birth
  Estimated gestational age (in days) of the child on the delivery date
Birthweight | Collected at time of birth
  Weight (in grams) of infant at birth

SECONDARY OUTCOMES:
Change in food spending | Baseline, around 3 months post-baseline, 60 days post-partum, one year post-partum
  A continuous measure asking about weekly expenditures on groceries and eating and restaurants, and other food options
Change in self reported physical and mental health | Baseline, around 3 months post-baseline, 60 days post-partum, one year post-partum
  Measures captured using an abbreviated 5-item Patient Reported Outcomes Measurement Information System (PROMIS) screener
Number of Prenatal Appointments | Collected quarterly from enrollment through birth
  Number of prenatal health appointments received during pregnancy
Maternal Immunizations Received | Collected quarterly from enrollment through birth
  Pregnancy-related immunizations received (e.g., Tdap, influenza) during pregnancy
Change in Maternal Platelet Count | Collected quarterly from enrollment through birth
  Change in lab results on platelet count from first prenatal visit to final prenatal visit
Change in Maternal White Blood Cell Count | Collected quarterly from enrollment through birth
  Change in lab results on while blood cell count from first prenatal visit to final prenatal visit
Change in Maternal Hematocrit Count | Collected quarterly from enrollment through birth
  Change in lab results on maternal hematocrit count from first prenatal visit to final prenatal visit
Change in Maternal Hemoglobin Count | Collected quarterly from enrollment through birth
  Change in lab results on maternal hemoglobin count from first prenatal visit to final prenatal visit
Change in Maternal Red Blood Cell Count | Collected quarterly from enrollment through birth
  Change in lab results on maternal red blood cell count from first prenatal visit to final prenatal visit
Maternal Anemia Diagnosis | Collected quarterly from enrollment through birth
  Incidence of maternal anemia diagnosis at any point during pregnancy
Fetal Complications Diagnosis | Collected quarterly from enrollment through birth
  Incidence of any common fetal complication diagnosis (e.g., ectopic pregnancy) at any point during pregnancy
Hypertensive Disorder Diagnosis | Collected quarterly from enrollment through birth
  Incidence of any hypertensive disorder diagnosis at any point during pregnancy
Spontaneous Preterm Labor | Collected quarterly from enrollment through birth
  Incidence of spontaneous preterm labor at any point during pregnancy
Preeclampsia Diagnosis | Collected quarterly from enrollment through birth
  Incidence of preeclampsia diagnosis at any point during pregnancy
Difficulty paying bills | Baseline, around 3 months post-baseline, 60 days post-partum, one year post-partum
  A single item measure capturing the incidence of bill payment difficulty in a typical month
Post-partum depression | Baseline, around 3 months post-baseline, 60 days post-partum, one year post-partum
  Collected through the Edinburgh Post-partum Depression Scale. This scale is score 0 to 30, with higher values indicator higher risk for post-partum depression
Intrauterine Fetal Demise (IUFD) | Collected quarterly from enrollment through birth
  Incidence of IUFD over course of pregnancy
Spontaneous Abortion | Collected quarterly from enrollment through birth
  Incidence of spontaneous abortion over course of pregnancy
Postpartum Complications | Birth through 60 days post-partum
  Incidence of common postpartum physical health complications (e.g., hypertension, sepsis)
Adverse Post-Partum Mental Health Diagnoses | Birth through 60 days post-partum
  Incidence of common postpartum adverse mental health diagnoses (e.g., anxiety, psychosis)
Maternal Mortality | Birth through 60 days post-partum
  Incidence of maternal mortality
Infant mortality | Birth through 60 days post-partum
  Incidence of infant mortality
Change in food quality | Baseline, around 3 months post-baseline, 60 days post-partum, one year post-partum
  A repeated assessment of the mix of foods consumed through the use of a 24-hour-recall-based food frequency questionnaire
Emergency liquidity | Baseline, around 3 months post-baseline, 60 days post-partum, one year post-partum
  A single item indicator capturing how participants would cover a $400 emergency expense
Public program participation | Baseline, around 3 months post-baseline, 60 days post-partum, one year post-partum
  A matrix question capturing the incidence of participation in common public welfare programs: Supplemental Nutrition Assistance (SNAP); Temporary Assistance for Needy Families (TANF); Public Housing/Housing Choice Vouchers; Women, Infants, and Children (WIC); Utility assistance; Child care assistance
Maternal Hospital Admissions | Collected quarterly from enrollment through one year post-partum
  Measure of hospital admissions derived from health care claims data
Maternal Emergency Room Visits | Collected quarterly from enrollment through one year post-partum
  Measure of emergency room visits derived from health care claims data
Maternal Wellness Visits | Collected quarterly from enrollment through one year post-partum
  Measure of wellness visits derived from health care claims data
Pediatric Visits | Birth through one year post-partum
  Number of pediatric visits in the post-partum period
Infant Adverse Health Diagnoses | Birth through one year post-partum
  Incidence of common infant adverse health diagnoses (e.g., colic, jaundice)
Days in Neonatal Intensive Care Unit (NICU) | Collected from birth through 60 days post-partum
  Length of NICU stay for infant following birth
Admission to Special Care Nursery | Collected from birth through 60 days post-partum
  Incidence of admission to special care nursery
Birth Defects | Collected from birth through 60 days post-partum
  Incidence of common birth defects (e.g., congenital heart defects, cleft palate)
Child Weight | Collected from birth through one year post-partum
  Child weight (grams) post-birth
Child Height | Collected from birth through one year post-partum
  Child height (centimeters) post-birth
Child Hospital Admissions | Collected from birth through one year post-partum
  Number of Hospital Admissions for Child Following Birth
Neonatal death | Collected from birth through one year post-partum
  Incidence of neonatal death
Child Emergency Department Admissions | Collected from birth through one year post-partum
  Number of emergency department admissions following birth

OTHER OUTCOMES:
Change in cooking skills | Baseline, around 3 months post-baseline, 60 days post-partum, one year post-partum
  Incidence of using basic and advanced kitchen tasks. Participants will be asked how often they perform an array of given tasks (Never, Rarely, Monthly, Weekly, Daily) such as boiling water, following a recipe, using a chef's knife, and so on, through a matrix question listing these tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Roll, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Operation Food Search Inc., St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No